CLINICAL TRIAL: NCT01711151
Title: Questionnaire Study for Patients With Interstitial Lung Disease
Brief Title: Interstitial Lung Disease Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 2012RESP05; UEAILDQUEST (Other: University of East Anglia)
Record Dates: First submitted 2012-10-09; First posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Interstitial Lung Disease
Keywords: ILD
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Idiopathic Pulmonary Fibrosis: Questionnaire evaluation
- Non Idiopathic Pulmonary Fibrosis: Questionnaire evaluation
- Sarciodosis: Questionnaire evaluation
- Healthy Controls: Questionnaire evaluation

SUMMARY:
1. To evaluate the health status of patients with Interstitial Lung Disease (ILD), and how this varies between subgroups of ILD.
2. To investigate the prevalence of symptoms, anxiety, depression, and sleep-disordered breathing within ILD patient population.
3. To assess the economic impact of ILD.
4. To understand how self-aware ILD patients are regarding their treatment/management.
5. To compare the demographic details, including smoking status and occupational history, of patients with interstitial lung disease

DETAILED DESCRIPTION:
Primary endpoint

• Health status in the target populations, as determined by the K-BILD questionnaire.

Secondary endpoints -

* Severity of dyspnoea suffered by patients
* Prevalence of anxiety and depression
* Prevalence of sleep-disordered breathing symptoms
* Degree of self-awareness displayed by patients
* The costs associated with ILD from a patient and healthcare perspective.
* Demographic details

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age greater than 18 years of age
* Any smoking status
* Diagnosis of Interstitial Lung Disease as defined below
* Full pulmonary lung function tests and routine immunological tests undertaken within 6 months of entry into study

Exclusion Criteria:

• Unable to give consent to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary Care
Sampling Method: Non-Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Difference in the Mean K-BILD score between the 4 groups | Baseline
  HRQL

SECONDARY OUTCOMES:
Severity of dyspnoea suffered by patients | Baseline
Prevalence of anxiety and depression | Baseline
Prevalence of sleep-disordered breathing symptoms | Baseline
Degree of self-awareness displayed by patients | Baseline
The costs associated with ILD from a patient and healthcare perspective | Baseline
Demographic details | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, Principal Investigator — University of East Anglia
Locations (1):
- Norfolk and Norwich Univeristy Hospital NHS foundation Trust, Norwich, Norfolk, United Kingdom